CLINICAL TRIAL: NCT01746498
Title: Therapeutic Effect of Direct Current Stimulation on Cognitive Function of Mild to Moderate Alzheimer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman M. Khedr, Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Direct current in Alzheimer's
Record Dates: First submitted 2012-11-30; First posted 2012-12-11 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer disease; Direct current stimulation; cognitive function; memory
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Active Comparator): 11 patients We Applied real anodal tDCS on the left dorsolateral prefrontal cortex (DLPFC)20 minutes every day for 10 consecutive days.
  Interventions: Procedure: Direct current stimulation using Anodal electrode
- Group 2 (Active Comparator): 11 patients we applied cathodal tDCS on left DLPFC for 20 minutes every day for 10 consecutive days.
  Interventions: Procedure: direct current stimulation using cathodal electrode
- Group 3 (Sham Comparator): 11 patients We applied sham stimulations(anodal tDCS) on the left DLPFC for few seconds the stop stimulations 2 mA every day for 10 days.
  Interventions: Procedure: Sham direct current stimulation

INTERVENTIONS:
Procedure: Direct current stimulation using Anodal electrode — 11 patients who received real anodal tDCS on the left DLPFC, 2 mA for 20 minute every day for 10 consecutive days
  Arms: Group 1
Procedure: direct current stimulation using cathodal electrode — 11 patients who received real cathodal tDCS on the left DLPFC, 2 mA for 20 minute every day for 10 consecutive days
  Arms: Group 2
Procedure: Sham direct current stimulation — 11 patients who received sham anodal tDCS on the left DLPFC just for few seconds, 2 ma, every day for 10 consecutive days
  Other Names: Direct current stimualtion (CX - 6650 Model TRCU - 04A Rolf Schneider Electronics, D-37130 Gleichen,; Germany).
  Arms: Group 3

SUMMARY:
The current study is planed to compare the efficacy of real (anodal and cathodal) vs sham transcranial direct current stimulation (tDCS) applied over the left dorsolateral prefrontal cortex (DLPFC) on cognitive functions and cortical excitability of patients with Alzheimer disease (AD).

Thirty three with mild to moderate Alzheimer's disease (AD) patients (diagnosis of probable AD according to the criteria of the National Institute of Neurological and Communicative Disorders and Stroke Alzheimer Disease and Related Disorders Association [NINCDS-ADRDA] were included in this study) were randomly classified into one of three groups (eleven for each group). The first group received anodal tDCS over left DLPFC and 2rd group received cathodal tDCS on the left DLPFC and the 3rd group received sham tDCS stimulation, daily for 10 consecutive days (5 days/week for 2 weeks). Minimental State Examination (MMSE), psychometric assessment for cognitive functions (MMSE, Wechsler memory scale, Wechsler adult Intelligent scale) were assessed before, after 10th sessions, and then after 1 and 2 month. Cortical excitability was assessed in both hemispheres before and after the end of sessions. Neurophysiological evaluations included resting and active motor threshold (rMT and aMT), and cortical silent period (CSP).

At the time of recruitment, none of the patients taking antidepressants, or neuroleptic, sedative-hypnotic drugs for at least two weeks before the assessment. All participants or their caregivers will give informed consent before participation in the test and after full explanation of the study protocol.

Outcome: The real group received (anodal and cathodal) tDCS are expected to have more improvement on cognitive functions compared to sham tDCS group. tDCS is considered new adjuvant non pharmacological therapeutic tool for management of AD patients with mild to moderate degree dementia.

ELIGIBILITY:
Inclusion Criteria:

* Thirty patients with a diagnosis of probable AD according to the criteria of the National Institute of Neurological and Communicative Disorders Association (NINCDS-ADRDA) (McKhann G et al.,1994) will be included in this study.

Exclusion Criteria:

* previous history of stroke
* Metabolic disturbances
* Other major medical illness or epilepsy
* Patients metallic objects in the body
* Patients subjected to a craniotomy in the past.

Ages: 45 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-06; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Minimental state Examination | base line and after 2 months
  To measure the cognitive function in alzheimer patients through measuring orientation, Registration, Attention and calculation, Recall,language, and copying with a total score 30.

SECONDARY OUTCOMES:
changes in cortical excitability | Base line and after 10 days
Wechsler memory scale | Basal and 2 months
Intelligent questant ( IQ) | basal and 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Eman Khedr, Asyut, Egypt